CLINICAL TRIAL: NCT01608490
Title: Lung Volume Reduction Coil Treatment in Patients With Emphysema (RENEW) Study
Acronym: RENEW
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA approval of supplementation to IDE to terminate subject long term follow up
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: PneumRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN0009
Record Dates: First submitted 2012-05-26; First posted 2012-05-31 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Emphysema
Keywords: COPD; RePneu
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: One group received standard of care and LVRC and the control group received only standard of care.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RePneu Lung Volume Reduction Coil System (Experimental): The RePneu Lung Volume Reduction Coil System is an implantable device, delivered through a fiber-optic bronchoscope. This is a two part system that consists of 1) sterile Nitinol Coils and 2) a sterile, disposable, single-use (single-patient) Delivery System consisting of a Guidewire, Catheter, Cartridge, and Forceps.
  Interventions: Device: RePneu Lung Volume Reduction Coil System
- Control arm is standard medical care (No Intervention): The Control Group will not undergo any bronchoscopies for Coil placement and will not receive prophylactic antibiotics or steroids before and after 'treatment' or chest x-rays in connection with the 'treatment' visits. The frequency of visits to the Study Doctor or designee will be similar to the LVRC Group.

INTERVENTIONS:
Device: RePneu Lung Volume Reduction Coil System — The LVRC group will undergo two bronchoscopic sessions under general or moderate sedation. During the procedure, subjects will be treated with Coils according to the Instructions for Use.
  Arms: RePneu Lung Volume Reduction Coil System

SUMMARY:
Multicenter, randomized, assessor-blinded controlled study of safety and effectiveness of the PneumRx, Inc. RePneu Lung Volume Reduction Coil (RePneu LVRC) System

DETAILED DESCRIPTION:
This will be a prospective, multicenter, randomized, assessor-blinded, controlled study comparing outcomes between the LVRC and Control Groups. Subjects will be block randomized in an LVRC (Treatment) to Control ratio of 1:1. The randomization will be stratified by homogeneous versus heterogeneous emphysema, to support a balance of patients with differing heterogeneity in both the LVRC and Control Groups.

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than or equal to 35 yrs of age
* CT Scan indicates bilateral emphysema, as determined by the Core Radiology Lab using the criteria presented in the "CT Scoring Plan for Core Radiology Lab"
* Subject has post-bronchodilator FEV1 less than or equal to 45% predicted
* Subject has Total Lung Capacity >100% predicted
* Subject has residual volume (RV) greater than or equal to 175% predicted
* Subject has marked dyspnea greater than or equal to 2 on mMRC scale of 0-4
* Subject has stopped smoking for at least 8 weeks prior to entering the study as confirmed by a Cotinine test or other appropriate diagnostic test.
* Subject has completed a pulmonary rehabilitation program within 6 mos prior to treatment and/or is regularly performing maintenance respiratory rehabilitation if initial supervised therapy occurred more than 6 mos prior to baseline testing.
* Subject has received Pneumococcal and Influenza vaccinations consistent with local recommendations and/or policy.
* Subject (and legal guardian, if applicable) has read, understood, and signed the Informed Consent form.

Exclusion Criteria:

* Subject has severe homogeneous emphysema determined by Core Radiology Lab.
* Subject has co-morbidities that may significantly reduce subject's ability to improve exercise capacity (e.g., severe arthritis, planned knee surgery) or baseline limitation on 6MWT is not due to dyspnea.
* Subject has a change in FEV1 of greater than 20% (or, for subjects with pre-bronchodilator FEV1 below 1L, a change of greater than 200mL) post-bronchodilator unless investigator can confirm by other means that subject does not have asthma.
* Subject has DLCO of less than 20% of predicted.
* Subject has severe gas exchange abnormalities, PaCO2 of greater than 55mm Hg; PaO2 of less than 45 mm Hg on room air (high altitude criterion: PaO2 of less than 30mm Hg).
* Subject has a history of recurrent clinically significant respiratory infections, defined as 3 hospitalizations for respiratory infection during the year prior to enrollment.
* Subject as severe pulmonary hypertension defined by right ventricular systolic pressure of greater than 50mm Hg via right heart catheterization and/or echocardiogram
* Subject has an inability to walk >140m (150 yd) in 6 minutes
* Subject has evidence of other severe disease (such as but not limited to lung cancer or renal failure), which in the judgment of the investigator may compromise survival of the subject for the duration of the study.
* Subject is pregnant or lactating, or plans to become pregnant within the study timeframe.
* Subject has an inability to tolerate bronchoscopy under moderate sedation or general anesthesia.
* Subject has clinically significant bronchiectasis.
* Subject has giant bullae >1/3 lung volume
* Subject has had previous LVR surgery, lung transplantation, lobectomy or LVR devices or other device to treat COPD in either lung.
* Subject has been involved in pulmonary drug or device studies within 30 days prior to this study.
* Subject is taking >20mg prednisone (or equivalent dose of a similar steroid) daily.
* Subject requires high level chronic immunomodulatory therapy to treat a moderate to severe chronic inflammatory autoimmune disorder.
* Subject is on an antiplatelet agent (such as Plavix) or anticoagulant therapy (such as Heparin or Coumadin) which cannot be stopped for 7 days prior to the procedure.
* Subject has any other disease, condition(s) or habit(s) that would interfere with completion of study and follow up assessments, would increase risks of bronchoscopy or assessments, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect study outcomes.
* Subject has a sensitivity or allergy to nitinol (nickel-titanium) or its constituent metals.
* Subject has a known sensitivity to drugs required to perform bronchoscopy.
* Subject has been diagnosed with alpha-1 antitrypsin deficiency (AATD).

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2019-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Strange, MD, Principal Investigator — Medical University of South Carolina
Locations (29):
- United States (23):
  - University of Alabama Lung Health Center, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - El Camino Hospital/Palo Alto Medical Foundation, Mountain View, California
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine - Yale New Haven Hospital, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Illinois Hospital and Health Center, Chicago, Illinois
  - Illinois Lung and Critical Care Institute, Peoria, Illinois
  - Pulmonary and Critical Care Associates of Baltimore, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - New York Presbyterian Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Temple, Philadelphia, Pennsylvania
  - Emphysema COPD Research Center, University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Pulmonary, Critical Care & Sleep Medicine Consultants,PCCS/St. Luke's Episcopal Hospital, Houston, Texas
  - University of Texas Health Sciences Center at San Antonio, San Antonio, Texas
  - Franciscan Research Center, Tacoma, Washington
  - University of Wisconsin School of Medicine & Public Health, Madison, Wisconsin
- Institut Universitaire de Cardiologie et de Pneumologie de Quebec (IUCPQ), Québec, Canada
- France (2):
  - Centre Hospitalier Universitaire de Nice, Nice
  - CHU de Reims - Hopital Maison Blanche, Reims
- Thoraxklinik University of Heidelberg, Heidelberg, Germany
- University Medical Center Groningen, Groningen, Netherlands
- Royal Brompton Hospital & Chelsea Westminster, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hartman JE, Shah PL, Sciurba F, Herth FJF, Slebos DJ; RENEW Study Group. Endobronchial coils for emphysema: Dual mechanism of action on lobar residual volume reduction. Respirology. 2020 Nov;25(11):1160-1166. doi: 10.1111/resp.13816. Epub 2020 Apr 8. PMID 32267059
- [Derived] Slebos DJ, Cicenia J, Sciurba FC, Criner GJ, Hartman JE, Garner J, Deslee G, Delage A, Jantz M, Marquette CH, Strange C, Hatipoglu U, Mehta AC, LaPrad AS, Schmid-Bindert G, Herth FJF, Shah PL; RENEW Study Group. Predictors of Response to Endobronchial Coil Therapy in Patients With Advanced Emphysema. Chest. 2019 May;155(5):928-937. doi: 10.1016/j.chest.2019.02.012. Epub 2019 Feb 21. PMID 30797746
- [Derived] Sciurba FC, Criner GJ, Strange C, Shah PL, Michaud G, Connolly TA, Deslee G, Tillis WP, Delage A, Marquette CH, Krishna G, Kalhan R, Ferguson JS, Jantz M, Maldonado F, McKenna R, Majid A, Rai N, Gay S, Dransfield MT, Angel L, Maxfield R, Herth FJ, Wahidi MM, Mehta A, Slebos DJ; RENEW Study Research Group. Effect of Endobronchial Coils vs Usual Care on Exercise Tolerance in Patients With Severe Emphysema: The RENEW Randomized Clinical Trial. JAMA. 2016 May 24-31;315(20):2178-89. doi: 10.1001/jama.2016.6261. PMID 27179849

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RePneu Lung Volume Reduction Coil System | Control Arm is Standard Medical Care
Started | 158 | 157
Completed | 141 | 142
Not Completed | 17 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RePneu Lung Volume Reduction Coil System | Control Arm is Standard Medical Care | Total
Number analyzed (Participants) | 158 | 157 | 315
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (8.05) | 64.3 (7.76) | 63.9 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 79 | 165
  Male | 72 | 78 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 157 | 155 | 312
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Meters: 6 Minute Walk Test - Change From Baseline to 12 Months Follow up
Description: mean absolute change from baseline at 12 months in the 6 Minute Walk Test comparing test and control groups (median if skewed)
Time Frame: baseline through 12 months follow up
Population: Patients who were analyzed at 12 months.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | RePneu Lung Volume Reduction Coil System | Control Arm is Standard Medical Care
Number analyzed (Participants) | 158 | 157
meters | 10.3 [-33.0 to 45.0] | -7.6 [-40.0 to 26.0]

2. Secondary Outcome: Mean Percent Change in FEV1 From Baseline to 12 Months
Description: Mean percent change in FEV1(Forced Expiratory Volume in 1 second) at 12 months (median if skewed)
Time Frame: BL to 12 months
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | RePneu Lung Volume Reduction Coil System | Control Arm is Standard Medical Care
Number analyzed (Participants) | 158 | 157
percentage change | 3.8 [-6.3 to 16.1] | -2.5 [-8.9 to 4.4]

3. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Mean Absolute Change From Baseline to 12 Months
Description: mean absolute difference in SGRQ results comparing BL to 12 months, LVRC vs. Control, score is on a scale from 0 to 100, negative change will be a better outcome.
Time Frame: BL to 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | RePneu Lung Volume Reduction Coil System | Control Arm is Standard Medical Care
Number analyzed (Participants) | 158 | 157
score on a scale | -8.1 (1.08) | 0.8 (1.05)

4. Secondary Outcome: 6MWT Responder Analysis
Description: 6MWT Responder Analysis: Responder is defined as those with an improvement of greater than or equal to 25 meters
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | RePneu Lung Volume Reduction Coil System | Control Arm is Standard Medical Care
Number analyzed (Participants) | 158 | 157
Participants | 60 | 41

5. Other Pre Specified Outcome: SGRQ Responder Analysis
Description: SGRQ Responder Analysis: Responder defined as those with an improvement greater than or equal to 4 points
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | RePneu Lung Volume Reduction Coil System | Control Arm is Standard Medical Care
Number analyzed (Participants) | 158 | 157
Participants | 98 | 48

6. Other Pre Specified Outcome: Residual Volume (RV) Mean Absolute Difference in RV From Baseline to 12 Months
Description: Mean absolute difference in RV results measured using plethysmography, comparing BL to 12 months, LVRC vs. Control
Time Frame: 12 months
Measure: Mean (Standard Error); unit: liters
Arm/Group | RePneu Lung Volume Reduction Coil System | Control Arm is Standard Medical Care
Number analyzed (Participants) | 158 | 157
liters | -0.41 (0.081) | -0.10 (0.080)

7. Other Pre Specified Outcome: RV/TLC Mean Absolute Difference From Baseline to 12 Months
Description: Mean absolute difference in RV/TLC (residual volume/total lung capacity - a measure done during lung function testing where residual volume is air left over in lung after completely breathing out and total lung capacity is how much air the lung can breathe in) results measured using plethysmography, comparing BL to 12 months, LVRC vs. Control
Time Frame: 12 months
Measure: Mean (Standard Error); unit: percent
Arm/Group | RePneu Lung Volume Reduction Coil System | Control Arm is Standard Medical Care
Number analyzed (Participants) | 158 | 157
percent | -3.96 (0.564) | -0.45 (0.554)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Complications occurring in the treatment arm were further categorized as device-related, procedure-related, or neither, and by those occurring during procedure hospitalization and those occurring post-discharge. Adverse events for the treatment group are only reported for subjects who began the treatment. Three (3) subjects discontinued the study prior to treatment, and are therefore not part of the safety population.
Arm/Group | RePneu Lung Volume Reduction Coil System | Control Arm is Standard Medical Care
All-Cause Mortality (participants affected / at risk) | 10/155 | 8/157
Serious Adverse Events (participants affected / at risk) | 78/155 | 44/157
Other Adverse Events (participants affected / at risk) | 155/155 | 142/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RePneu Lung Volume Reduction Coil System (N=155) | Control Arm is Standard Medical Care (N=157)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 5 (5) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy to metals (Immune system disorders) | 1 (1) | 0 (0)
Latex allergy (Immune system disorders) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 5 (5) | 2 (2)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 3 (3) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Lung infection (Infections and infestations) | 2 (3) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 31 (34) | 8 (10)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Subacute endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Influenza A virus test positive (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign lymph node neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 43 (70) | 32 (46)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Coeliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Haemotoma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RePneu Lung Volume Reduction Coil System (N=155) | Control Arm is Standard Medical Care (N=157)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhthmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 4 (5)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 3 (3)
Cataract (Eye disorders) | 1 (1) | 3 (3)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth fracture (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 3 (3) | 0 (0)
Chest discomfort (General disorders) | 20 (30) | 1 (1)
Chest pain (General disorders) | 10 (14) | 4 (4)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 3 (3) | 0 (0)
Injection site extravasation (General disorders) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 7 (8) | 0 (0)
Medical device pain (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 21 (28) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 11 (11) | 4 (4)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy to metals (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Latex allergy (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 2 (2)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (2) | 2 (2)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 21 (31) | 25 (32)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 4 (4) | 0 (0)
Candidiasis (Infections and infestations) | 5 (5) | 3 (4)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 2 (3)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Ersipelas (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Genital abscess (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Infected bites (Infections and infestations) | 0 (0) | 1 (1)
Infectious disease carrier (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 5 (5) | 3 (3)
Laryngitis fungal (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 2 (4) | 2 (2)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 10 (13) | 6 (6)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 10 (13) | 4 (6)
Oral fungal infection (Infections and infestations) | 1 (2) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 36 (44) | 12 (14)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory monoliasis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2)
Rhinitis (Infections and infestations) | 2 (2) | 5 (5)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4) | 8 (12)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Sputum purulent (Infections and infestations) | 1 (1) | 2 (2)
Subacute endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (2)
Tracheobronchitis (Infections and infestations) | 3 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 9 (9)
Urinary tract infection (Infections and infestations) | 5 (8) | 6 (6)
Volvovaginal mycotic infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Antibiotic resistant Staphylococcus test positive (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0)
Influenza A virus test positive (Investigations) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Sputum abnormal (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Overweight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 18 (23) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 3 (3)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (4)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 4 (5)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 1 (1)
Somnambulism (Psychiatric disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 6 (6) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 108 (228) | 91 (185)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (41) | 3 (3)
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 (41) | 12 (15)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 91 (140) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (16) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sputum discolored (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 14 (22) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sinus operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Coeliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Haemotoma (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 2 (2)
Hypotension (Vascular disorders) | 6 (7) | 0 (0)
Phlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Venous insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Genital Herpes (Infections and infestations) | 1 (1) | 0 (0)
Benign Lymph Node Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No